CLINICAL TRIAL: NCT06717243
Title: A Prospective Observational Study on Genomic and Methylation Signatures in Patients with Extensive-Stage Small Cell Lung Cancer and Metastatic Large Cell Neuroendocrine Carcinoma Undergoing Chemo-Immunotherapy
Brief Title: Genomic and Methylation Markers in SCLC and LCNEC for Chemo-Immunotherapy Resistance Prediction (STRATUS)
Acronym: STRATUS
Status: Recruiting | Type: Observational
Sponsor: Oncology Center of Biochemical Education And Research (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Icahn School of Medicine at Mount Sinai (Other); Sotiria General Hospital (Other)
Responsible Party: Principal Investigator, Kostas N.Syrigos, Professor of Medicine and Medical Oncology, Oncology Center of Biochemical Education And Research
Other Study IDs: 2082/19-01-2024
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Small Cell Lung Cancer; Large Cell Neuroendocrine (NE) Tumors; Treatment Failure; Biomarkers / Blood; Biomarkers; Immunotherapy
Keywords: Small Cell Lung Cancer (SCLC); Large Cell Neuroendocrine Carcinoma (LCNEC); Chemo-Immunotherapy; Treatment Resistance; Circulating Tumor Cells (CTCs); Circulating Tumor DNA (ctDNA); Liquid Biopsy; Genomic Profiling; Epigenetics; Biomarker Discovery; Lung Cancer; Molecular Signatures; Clonal Evolution; Personalized Oncology; Cancer Immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms; Neoplastic Cells, Circulating; Lung Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will retain the following types of biospecimens:
  Blood samples: Plasma, serum, and buffy coat for analysis of circulating tumor DNA (ctDNA), circulating tumor cells (CTCs), and other molecular markers.
  Tumor tissue samples: Fresh-frozen and formalin-fixed paraffin-embedded (FFPE) tumor biopsies for genomic, epigenetic, and transcriptomic analyses.
  Optional re-biopsy samples: Collected from newly emerged lesions during disease progression to study clonal evolution and resistance mechanisms.
  All samples will be securely stored in a biorepository, de-identified, and used for DNA extraction and molecular profiling, including next-generation sequencing and DNA methylation analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Extensive-Stage Small Cell Lung Cancer (ES-SCLC) patients: This cohort includes adults with extensive-stage small cell lung cancer (ES-SCLC) receiving standard-of-care chemo-immunotherapy, such as platinum-based chemotherapy (cisplatin or carboplatin) combined with immune checkpoint inhibitors (atezolizumab or durvalumab). The study collects biospecimens, including blood (for circulating tumor DNA and circulating tumor cells) and tumor tissue, at baseline, during treatment, and at progression. These samples are analyzed to identify genomic, epigenetic, and transcriptomic signatures associated with treatment resistance. Insights gained will improve understanding of resistance mechanisms and guide personalized treatment strategies for ES-SCLC.
  Interventions: Drug: Carboplatin/Cisplatin -Etoposide - Atezolizumab
- Large Cell Neuroendocrine Carcinoma (LCNEC) patients: This cohort includes adults diagnosed with metastatic large cell neuroendocrine carcinoma (LCNEC). Participants will receive standard-of-care systemic therapies, such as platinum-based chemotherapy (cisplatin or carboplatin), with or without immune checkpoint inhibitors, based on physician discretion.
  Biospecimens, including blood (for circulating tumor DNA and circulating tumor cells) and tumor tissue, will be collected at baseline, during treatment, and upon disease progression. These samples will undergo molecular analysis to identify genomic, epigenetic, and transcriptomic changes associated with treatment resistance and progression.
  Interventions: Drug: Carboplatin/Cisplatin -Etoposide - Atezolizumab

INTERVENTIONS:
Drug: Carboplatin/Cisplatin -Etoposide - Atezolizumab — This intervention represents the standard-of-care first-line treatment regimen for extensive-stage small cell lung cancer (ES-SCLC). The regimen includes:
  Carboplatin or Cisplatin: Platinum-based chemotherapeutic agents that cause DNA cross-linking, leading to tumor cell death.
  Etoposide: A topoisomerase II inhibitor that prevents DNA replication and tumor growth.
  Atezolizumab: A PD-L1 immune checkpoint inhibitor that enhances the immune system's ability to detect and destroy cancer cells.
  This combination therapy is administered as part of routine clinical practice. The study does not investigate the efficacy or safety of these drugs but rather focuses on analyzing molecular changes in tumors, such as genomic and epigenetic alterations, to understand mechanisms of treatment resistance. Biospecimens are collected from patients during treatment and progression for detailed analysis.

SUMMARY:
The goal of this observational study is to understand how genomic and epigenetic factors contribute to resistance against chemo-immunotherapy in adults diagnosed with extensive-stage small cell lung cancer (ES-SCLC) or metastatic large cell neuroendocrine carcinoma (LCNEC). Both ES-SCLC and LCNEC are aggressive forms of lung cancer with limited treatment options and poor prognosis. While initial responses to chemo-immunotherapy are often promising, most patients develop resistance within a few months, resulting in disease progression and limited survival. This study seeks to explore the molecular and cellular changes that drive resistance, providing insights that could guide more personalized and effective treatment strategies in the future.

The study focuses on identifying genomic and methylation signatures, as well as analyzing circulating tumor cells (CTCs) and tumor DNA (ctDNA), to better understand the mechanisms of resistance. By collecting and analyzing these biomarkers over time, researchers aim to identify patterns that distinguish patients who benefit long-term from therapy from those who experience early resistance. These findings may pave the way for new diagnostic tools and therapies to predict and overcome resistance to chemo-immunotherapy.

The main questions this study seeks to answer are:

Are there specific genomic or methylation patterns that predict resistance to chemo-immunotherapy in ES-SCLC and LCNEC? How are circulating tumor cells (CTCs) and tumor DNA (ctDNA) associated with disease progression, treatment response, and survival? What molecular differences exist between patients who respond long-term and those who develop resistance early in their treatment?

Participants will:

Provide blood and tumor tissue samples before treatment to establish baseline molecular profiles.

Undergo follow-up visits every 9 weeks during treatment, where additional blood samples and imaging tests will be collected to monitor disease progression and treatment response.

Optionally provide tissue samples through re-biopsy if the disease progresses, enabling researchers to compare changes in tumor biology over time.

All blood and tissue samples will be de-identified and securely stored for genomic and epigenetic analyses. Blood samples will be examined for circulating tumor cells and tumor DNA, while tumor tissue samples will undergo in-depth genomic and methylation profiling. Researchers will use advanced molecular and bioinformatics techniques to uncover specific patterns associated with resistance, aiming to improve current treatment strategies and develop more precise therapies.

The study will analyze data from patients over three years, encompassing various stages of treatment and disease progression. By examining longitudinal samples, the study aims to capture the dynamic changes that occur in the tumor microenvironment and how these relate to treatment outcomes.

This research is particularly important because current treatment options for ES-SCLC and LCNEC are limited, and there are no established methods to predict which patients will respond to chemo-immunotherapy. Identifying biomarkers of resistance could transform clinical care, allowing oncologists to tailor treatments to individual patients' molecular profiles and improve survival outcomes.

Ultimately, the findings from this study could lead to the development of new biomarkers for resistance, improve early detection of treatment failure, and provide the foundation for novel therapies targeting resistant cancer cells. By addressing a critical gap in the understanding of resistance mechanisms, the STRATUS trial has the potential to significantly advance the field of personalized oncology.

DETAILED DESCRIPTION:
The STRATUS Trial (Study of Tumor Characteristics and Molecular Signatures in Neuroendocrine Tumors and SCLC) is an ambitious, prospective observational study designed to explore the molecular and genomic mechanisms underlying resistance to chemo-immunotherapy in patients diagnosed with extensive-stage small cell lung cancer (ES-SCLC) and metastatic large cell neuroendocrine carcinoma (LCNEC). These two aggressive forms of cancer represent a significant unmet clinical need, with high relapse rates and limited therapeutic options available following the development of treatment resistance.

The study seeks to uncover actionable biomarkers, characterize resistance mechanisms, and improve our understanding of tumor evolution under selective pressures from standard therapies. By leveraging cutting-edge molecular techniques, such as next-generation sequencing (NGS), DNA methylation profiling, and liquid biopsies, STRATUS aims to set the foundation for personalized cancer treatment approaches in these difficult-to-treat malignancies.

Background and Rationale The Challenge of Resistance in ES-SCLC and LCNEC Small cell lung cancer (SCLC) and large cell neuroendocrine carcinoma (LCNEC) are both high-grade neuroendocrine tumors characterized by rapid growth, early dissemination, and a poor prognosis. Approximately two-thirds of SCLC cases are diagnosed as extensive-stage disease (ES-SCLC), where the tumor has spread beyond the hemithorax and regional lymph nodes. Similarly, LCNEC, though rare, is frequently diagnosed at metastatic stages, with limited systemic treatment options available.

Standard treatment for ES-SCLC includes platinum-based chemotherapy combined with immune checkpoint inhibitors (ICIs), such as atezolizumab or durvalumab. While initial response rates exceed 70%, resistance develops rapidly in most patients, leading to disease progression within months. For LCNEC, the therapeutic landscape is even more limited, with a lack of targeted therapies or predictive biomarkers guiding treatment.

Need for Molecular Insights Resistance mechanisms in these cancers are thought to involve tumor heterogeneity, clonal evolution, epigenetic modifications, and immune evasion. However, the exact processes that drive resistance remain poorly characterized. Molecular profiling offers an opportunity to identify genomic and epigenetic alterations that correlate with treatment failure, allowing for the development of predictive biomarkers and targeted therapeutic strategies.

Role of Liquid Biopsies Liquid biopsies, including the analysis of circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA), have emerged as powerful tools for non-invasive tumor monitoring. These biomarkers provide real-time insights into tumor dynamics, enabling the detection of resistance mechanisms, clonal evolution, and molecular relapse.

Study Objectives Primary Objective To identify and characterize genomic, epigenetic, and methylation signatures associated with resistance to chemo-immunotherapy in ES-SCLC and LCNEC patients.

Secondary Objectives To evaluate the relationship between circulating biomarkers (CTCs, ctDNA) and clinical outcomes, including progression-free survival (PFS) and overall survival (OS).

To compare molecular profiles between long-term responders and patients who develop early resistance.

To assess tumor-immune interactions and their role in resistance mechanisms, focusing on PD-L1 expression, T-cell exhaustion, and cytokine signaling pathways.

Exploratory Objectives To investigate clonal evolution and emergent subpopulations associated with resistance using phylogenetic analyses.

To explore spatial transcriptomic patterns within the tumor microenvironment. To evaluate the potential of novel biomarkers for guiding treatment decisions and monitoring disease progression.

Study Design The STRATUS Trial is a multicenter, prospective observational study involving patients treated at the 3rd Department of Medicine, National and Kapodistrian University of Athens, Sotiria Hospital, and other participating centers. The study includes detailed clinical, molecular, and imaging assessments over a three-year follow-up period.

Inclusion Criteria Adults aged 18-85 years diagnosed with ES-SCLC or LCNEC. ECOG performance status of 0-2. Histological confirmation of diagnosis with available tumor tissue for molecular analysis.

At least one measurable or evaluable lesion according to RECIST 1.1 criteria. Willingness to provide blood samples and participate in follow-up visits. Exclusion Criteria Inability to tolerate chemo-immunotherapy. Presence of another active malignancy or significant comorbidity. Patients with no measurable disease or inadequate follow-up potential. Data Collection and Sample Handling Baseline Assessments

Before starting treatment, participants will undergo:

Comprehensive clinical evaluations, including medical history, ECOG performance status, and comorbid conditions.

Imaging studies (e.g., CT, PET) to assess tumor burden and metastatic sites. Blood sample collection for baseline ctDNA and CTC analysis. Tumor biopsies for genomic, transcriptomic, and methylation profiling. On-Treatment Monitoring

Participants will attend follow-up visits every 9 weeks, during which:

Blood samples will be collected to monitor ctDNA and CTC levels. Imaging studies will evaluate tumor response according to RECIST 1.1 criteria. Adverse events, clinical progression, and treatment modifications will be documented.

Disease Progression Assessments

For patients with progressive disease:

Repeat biopsies of newly emerging lesions will be performed to identify resistance-associated changes.

Blood samples will capture dynamic shifts in ctDNA and CTC profiles, enabling comparisons with baseline and on-treatment data.

Laboratory Methods NGS-Based Genomic Analysis: Comprehensive sequencing will identify mutations, copy number alterations, and structural rearrangements.

Epigenetic Profiling: DNA methylation arrays will uncover resistance-related epigenetic changes.

Spatial Transcriptomics: High-resolution analysis of tumor microenvironment architecture and gene expression patterns.

Statistical Analysis Sample Size A total of 111 patients will be enrolled, providing sufficient power to detect significant differences in molecular markers across subgroups.

Primary Analysis Regression models will evaluate associations between molecular markers and treatment resistance.

Descriptive statistics will summarize biomarker distributions and clinical outcomes.

Secondary Analysis Kaplan-Meier survival curves will estimate PFS and OS. Cox proportional hazards models will assess the prognostic significance of identified biomarkers.

Exploratory Analysis Machine learning models will predict resistance based on integrated multi-omic data.

Clonal evolution will be modeled using phylogenetic techniques to trace tumor adaptation under therapeutic pressure.

Ethical Considerations The study will comply with the Declaration of Helsinki and GDPR guidelines for data protection. Participants will provide written informed consent, and all data will be de-identified to ensure confidentiality.

Significance and Anticipated Impact

The STRATUS Trial is expected to:

Identify actionable biomarkers for predicting and overcoming resistance. Advance the understanding of tumor evolution and immune evasion in SCLC and LCNEC.

Guide the development of personalized treatment strategies, ultimately improving patient outcomes.

Conclusion The STRATUS Trial represents a landmark effort to address the challenges of resistance in SCLC and LCNEC. By combining advanced molecular analyses with robust clinical monitoring, this study has the potential to transform the management of these aggressive cancers and pave the way for a new era of precision oncology.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 18-85 years.
* Histologically confirmed locally advanced extensive-stage small cell lung cancer (ES-SCLC).
* Histologically confirmed locally advanced or metastatic large cell neuroendocrine carcinoma (LCNEC).
* Treatment Plan: Eligible patients must be initiating standard-of-care chemo-immunotherapy, including platinum-based chemotherapy (cisplatin or carboplatin) combined with immune checkpoint inhibitors (atezolizumab or durvalumab).
* Measurable Disease: At least one measurable or evaluable lesion as defined by RECIST 1.1 criteria.
* Baseline Biospecimen Availability: Patients must agree to provide baseline blood and tumor biopsy samples for molecular and genomic analyses.
* Treatment Naïve for Study Indication: Patients should not have received prior systemic therapy for ES-SCLC or LCNEC.
* Life Expectancy: Estimated life expectancy of at least 3 months, as determined by the treating physician.
* Follow-Up Commitment: Willingness to attend scheduled follow-up visits and provide additional biospecimens (blood and/or tissue) during treatment and at progression.
* Performance Status: ECOG performance status of 0-2.
* Organ Function: Adequate hematologic, renal, and hepatic function as per the treating physician's discretion.
* Consent: Ability and willingness to provide written informed consent for participation in the study and collection of biospecimens (e.g., blood and tumor tissue).
* Compliance with Study Protocol: Demonstrated ability and willingness to comply with all study-related procedures, including biospecimen collection and follow-up visits.
* Non-Pregnant and Non-Lactating: Women of childbearing potential must have a negative pregnancy test at baseline and agree to use effective contraception during the study period.
* Immunotherapy Eligibility: Patients must not have contraindications to immune checkpoint inhibitors (e.g., autoimmune diseases requiring systemic immunosuppressive therapy).
* Platinum-Based Therapy Tolerance: Patients must be deemed medically fit to receive platinum-based chemotherapy (cisplatin or carboplatin) as determined by the treating physician.
* No Active Infections: Patients must not have active, uncontrolled infections, including but not limited to tuberculosis, hepatitis B, hepatitis C, or HIV.
* Psychosocial Stability: Patients must have adequate psychosocial support and the mental capacity to understand and provide informed consent for participation in the study.
* Stable Brain Metastases: Patients with brain metastases are eligible if the metastases have been treated (e.g., surgery or radiotherapy) and are stable for at least 4 weeks prior to enrollment, as confirmed by imaging.
* Steroid Use for Brain Metastases: Patients requiring corticosteroids for brain metastases are eligible only if they are on a stable or tapering dose equivalent to ≤10 mg/day of prednisone for at least 2 weeks prior to enrollment.

Exclusion Criteria:

* Uncontrolled Brain Metastases: Patients with untreated or progressive brain metastases causing significant neurological symptoms.
* Concurrent Malignancies: Presence of any active malignancy other than ES-SCLC or LCNEC within the past 3 years, except for treated non-melanoma skin cancer or in situ cervical carcinoma.
* Previous Systemic Therapy: Prior systemic chemotherapy or immunotherapy for ES-SCLC or LCNEC.
* Severe Comorbidities: Significant comorbidities, such as uncontrolled cardiovascular, respiratory, or autoimmune diseases, that could interfere with study participation or treatment.
* Active Infection: Patients with active infections requiring systemic therapy, including tuberculosis, hepatitis B or C, or HIV.
* Pregnancy or Lactation: Pregnant or lactating women, or women of childbearing potential who are not using effective contraception.
* Immunosuppressive Therapy: Patients requiring systemic immunosuppressive therapy, including high-dose corticosteroids (equivalent to >10 mg/day prednisone), within 2 weeks prior to enrollment.
* Severe Allergic Reactions: History of severe hypersensitivity reactions to any component of the planned treatment regimen, including platinum-based chemotherapy or immune checkpoint inhibitors.
* Life-Threatening Conditions: Life expectancy less than 3 months, as assessed by the treating physician.
* Inability to Comply: Patients unable or unwilling to adhere to study protocols, including biospecimen collection and follow-up visits.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 18 to 85 years diagnosed with extensive-stage small cell lung cancer (ES-SCLC) or metastatic large cell neuroendocrine carcinoma (LCNEC). Participants must have histologically confirmed disease and at least one measurable lesion as per RECIST 1.1 criteria. Eligible patients are those initiating standard-of-care chemo-immunotherapy, including platinum-based chemotherapy (cisplatin or carboplatin) combined with immune checkpoint inhibitors (atezolizumab or durvalumab). Patients with ECOG performance status of 0-2 and adequate organ function are included. Exclusion criteria involve prior systemic therapy for ES-SCLC or LCNEC, concurrent malignancies, or severe comorbidities. The study population will provide blood and tumor tissue samples for molecular analyses, aiming to uncover resistance mechanisms and develop predictive biomarkers for treatment outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Genomic and Epigenetic Alterations Associated with Resistance to Chemo-Immunotherapy | Baseline to disease progression (up to 36 months).
  Identification of genomic, methylation, and other epigenetic alterations that are associated with resistance to standard-of-care chemo-immunotherapy (platinum-based chemotherapy combined with immune checkpoint inhibitors) in patients with extensive-stage small cell lung cancer (ES-SCLC) and metastatic large cell neuroendocrine carcinoma (LCNEC).

SECONDARY OUTCOMES:
Association Between Circulating Biomarkers and Clinical Outcomes (PFS, OS) in Chemo-Immunotherapy Recipients | Baseline to 36 months.
  Evaluation of the correlation between circulating tumor cells (CTCs), circulating tumor DNA (ctDNA), and clinical outcomes, including progression-free survival (PFS) and overall survival (OS), in patients receiving chemo-immunotherapy for extensive-stage small cell lung cancer (ES-SCLC) and metastatic large cell neuroendocrine carcinoma (LCNEC).

OTHER OUTCOMES:
Molecular Changes in Tumor Microenvironment and Immune Response | Baseline to disease progression (up to 36 months).
  Characterize changes in the tumor microenvironment (TME), including immune cell infiltration, PD-L1 expression, and cytokine signaling, during and after chemo-immunotherapy in patients with ES-SCLC and LCNEC.

CONTACTS AND LOCATIONS:
Locations (2):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- 3rd Department of Medicine, National and Kapodistrian University of Athens, Sotiria Hospital, Athens, Greece